CLINICAL TRIAL: NCT01132300
Title: An Open Trial Evaluating Efficacy of NeMa-st - A Computerized, Image Guided, Auto-Targeted Neurostimulation Device for the Treatment of Non Specific Low Back Pain
Brief Title: Efficacy Study Image Guided, Auto-Targeted Neurostimulation for the Treatment of Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Nervomatrix Ltd. Israel (Unknown)
Responsible Party: Elad Schiff, MD, Bnai Zion Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Approval Pending
Record Dates: First submitted 2009-09-15; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Image Guided TENS (Auto-Targeted Neurostimulation, NeMa-st)

INTERVENTIONS:
Device: Image Guided TENS (Auto-Targeted Neurostimulation, NeMa-st) — Patients will undergo 2 treatments per week during 4 weeks using the device. During the study Patients are allowed to maintain/continue taking medications/ analgesics for pain relief prescribed to them before the study. Medication use will be recorded.
  Other Names: Nervomatrix Ltd. Auto-Targeted Neurostimulation, NeMa-st

SUMMARY:
The purpose of this study is:

* Initial evaluation of the clinical effectiveness of Image Guided Transcutaneous Electrical Stimulation (TENS) device for treatment of non-specific low back pain.
* To assess the tolerability and acceptability of the device by the caregiver ("User Friendly").
* To evaluate patients' tolerance by monitoring side effects and tolerability during treatment.

DETAILED DESCRIPTION:
Transcutaneous electrical nerves stimulation (TENS) devices are a drug-free alternative for managing pain. For the past thirty years, doctors have been prescribing FDA approved TENS worldwide as an effective way to relieve pain. TENS device currently utilized includes a variety of types of devices and pulse modulations. Most of these devices are applied on large surface areas, and are designed to block the pain signal (gate mechanism) to the brain. Others manual TENS devices are applied to small surface areas to stimulate peripheral nerve ends, and by that causing the release of endorphins with a significantly superior clinical outcome. Such treatments are time consuming and cumbersome and requires previous knowledge of location of nerve ends.

A novel device capable of scanning a large skin surface area, automatically locating nerve ends responsible for pain relief by utilizing skin impedance measurements and image processing with anatomical matching will be tested for stimulating these peripheral nerve ends (NeMa-st, Nervomatrix Ltd., Netanya, Israel).

For this purpose an open study to initially evaluate safety and efficacy of the intervention is designed. 20 patients will undergo 2 treatment sessions per week for a period of 4 weeks, while maintaining their pain relief medication treatment regime.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific low back pain persisted at least 1 month and no longer than 12 month before the study
* Patients must have a baseline score>40 mm on the VAS pain scale
* If taking analgesics, patients must agree to maintain a steady regimen for the duration of the study.
* Able to provide written and verbal informed consent.

Exclusion Criteria:

* Sciatica
* Diagnosed spinal stenosis
* Back Pain potentially attributable to specific underlying diseases or conditions (e.g. pregnancy, metastatic cancer, spondylolisthesis, fractured bones, dislocated joints, disc eruption).
* Unstable medical or severe psychiatric conditions or dementia.
* Previous Back surgery
* Physically unable to undergo treatment
* Patients receiving workers compensation or those involved in litigation
* Minimal pain - less than 40mm score on VAS scale
* History of pacemaker , implantable devices, history of cardiac arrhythmias
* Allergy or intolerance to adhesive materials
* Clinical evidence of cardiovascular, pulmonary, renal, hepatic, neurological , hematological or endocrine abnormalities.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale Pain Questionnaire (VAS) | Baseline, before, and two hours after treatment session, 2 times a week, up to 5 weeks

SECONDARY OUTCOMES:
Oswestry Disability Questionnaire | once a week during the study, up to 5 weeks
Side effect record | after each treatment session, 2 times a week, up to 5 weeks
Range of Motion - lower back and pelvic forward flexion | Baseline, once a week, up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elad Schiff, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel